CLINICAL TRIAL: NCT02546830
Title: Automatic Oxygen Administration in Early and Late Postoperative Hypoxaemia Prevention After Major Abdominal and Thoracic Surgery
Brief Title: Automatic Oxygen Administration After Major Abdominal and Thoracic Surgery
Acronym: FreeO2PostOp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RB14-060; CHRU de Brest (Registry Identifier: RB14-060)
Record Dates: First submitted 2015-08-20; First posted 2015-09-11 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Major Thoracic and Abdominal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FreeO2 v2.2 active (Experimental): Automatic Oxygen Administration
  Interventions: Device: FreeO2 v2.2 active
- FreeO2 v2.2 with manual oxygenation (Active Comparator): Manual Oxygen Administration
  Interventions: Device: FreeO2 v2.2 with manual oxygenation

INTERVENTIONS:
Device: FreeO2 v2.2 active — * Automatic adjustment of oxygen through the "Free O2" device.
  * "FreeO2" device in mode medical data collecting(SpO2,EtCO2...).
  Arms: FreeO2 v2.2 active
Device: FreeO2 v2.2 with manual oxygenation — * Manual adjustment of oxygen without the assistance of the "FreeO2" device.
  * Only "FreeO2" device in mode medical data collecting(SpO2,EtCO2...).
  Arms: FreeO2 v2.2 with manual oxygenation

SUMMARY:
The aim of the study is to assess the use feasibility of the FreeO2 system so as to deliver automatically oxygen in the post anesthesia care unit in a patient population admitted for major abdominal and thoracic surgery.

The investigators' hypothesis is that FreeO2 system will provide a better control of the oxygen saturation and reduce postoperative hypoxaemia.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative anesthetic visit for major thoracic or abdominal surgery ( ARISCAT risk score ≥ 26) with general anesthesia
* Patient consent

Randomization Criteria:

* Admission in post-anesthesia care unit after major thoracic or abdominal surgery
* Randomization and device establishment within a time less than one hour after the endotracheal intubation
* Availability of the prototype FreeO2
* Absence of criteria of gravity justifying immediately a different technique of ventilatory support:

  * Disturbance of consciousness with a Glasgow Coma Score ≤ 12
  * Serious ventricular rhythm disorders
  * Hemodynamic instability (SBP <80mmHg or recourse to vasopressors)
  * Cardiac or respiratory arrest
  * pH < 7.35 and PaCO2 > 55 mm Hg
* Necessity of an oxygen flow less than 15 L / min to maintain a SpO2 higher than 92%.
* Absence of necessity of a urgent surgery
* Oxygen saturation measured by Spo2 sensor

Exclusion Criteria:

* BMI ≥ 35 kg/m2
* Obstructive sleep Apnea (with or without Mechanical therapy)
* Emergency Surgery for life-threatening
* Age <18 years
* Pregnant women, lactating
* perturbed or non-cooperative patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in the target zone of oxygen saturation | 3 days
  The target zone of oxygen saturation is : SpO2 = 88-92% for COPD patient and 92-96% for non COPD

SECONDARY OUTCOMES:
nursing workload | 3 days
  nursing workload assessed by the number of manual Oxygen flow adjustments and airway management procedures
Time spent in a area of severe desaturation (SpO2 <85%) | 3 days
  Time spent in a area of severe desaturation (SpO2 <85%) evaluated by freeO2 device
Time spent in a hyperoxia area (SpO2> 98%). | 3 days
  Time spent in a hyperoxia area (SpO2> 98%) evaluated by freeO2 device
Maintaining EtCO2 in a selected area | 3 days
  Maintaining EtCO2 in a selected area evaluated by freeO2 device
Oxygen consumption measured at the end of administration | 3 days
  Oxygen consumption measured at the end of administration
Duration of oxygen administration during hospitalization | 3 days
  Duration of oxygen administration during hospitalization
Number of complications related to the administration of oxygen | 28 days max
  Number of complications related to the administration of oxygen
Frequency of use of ventilation (invasive or noninvasive ) | 28 days max
  Frequency of use of ventilation (invasive or noninvasive )
Duration of hospitalization | 28 days max
  Duration of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Erwan L'HER, Principal Investigator — University Hospital, Brest
Locations (5):
- Hôpital Laval - Québéc, Québéc, Canada
- France (4):
  - Brest, University Hospital, Brest
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Montpellier, Montpellier
  - CHU Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] L'Her E, Jaber S, Verzilli D, Jacob C, Huiban B, Futier E, Kerforne T, Pateau V, Bouchard PA, Consigny M, Lellouche F. Automated closed-loop versus standard manual oxygen administration after major abdominal or thoracic surgery: an international multicentre randomised controlled study. Eur Respir J. 2021 Jan 5;57(1):2000182. doi: 10.1183/13993003.00182-2020. Print 2021 Jan. PMID 32855218
- [Derived] L'her E, Jaber S, Verzilli D, Jacob C, Huiban B, Futier E, Kerforne T, Pateau V, Bouchard PA, Gouillou M, Nowak E, Lellouche F. Automated oxygen administration versus conventional oxygen therapy after major abdominal or thoracic surgery: study protocol for an international multicentre randomised controlled study. BMJ Open. 2019 Jan 17;9(1):e023833. doi: 10.1136/bmjopen-2018-023833. PMID 30782716